CLINICAL TRIAL: NCT02469571
Title: Modulation of Gut Microbiota in Early Sepsis: A Pilot Study
Acronym: MGM-sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 26-496 ex 13/14
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): 5 g of Winclove-607 containing Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Enterococcus faecium W54, Lactobacillus acidophilus W37, Lactobacillus acidophilus W55, Lactobacillus paracasei W20, Lactobacillus plantarum W1, Lactobacillus plantarum W62, Lactobacillus rhamnosus W71, Lactobacillus salivarius W24 at a concentration of 1.1 x 109 cfu/g twice daily for the 4 weeks
  Interventions: Dietary Supplement: Winclove 607
- Placebo (Placebo Comparator): a similar looking and tasting placebo without bacteria once daily for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Winclove 607 — multispecies probiotic
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Background Sepsis is a common disease leading to high morbidity and mortality. Gut microbiota and/or gut permeability may play a crucial role in the development of organ dysfunction.

Hypothesis The ingestion of a multispecies probiotic in early sepsis is able to modulate gut microbiota and/or gut permeability.

DETAILED DESCRIPTION:
Sepsis is a systemic deleterious host response to infection causing major healthcare problems. Sepsis affects millions of people around the world each year, with a lethality of 25%-50%. The incidence is increasing partly because of a raise in average age and occurrence of predisposing diseases in the population, and partly because of shifts in causative pathogens. Effectiveness of therapy administered in the initial hours of severe sepsis critically influences the clinical outcome of the patient.

Lacking reliable biomarkers for early stages, the diagnosis of (severe) sepsis relies on a combination of surrogate parameters indicating end organ dysfunction.

Recently, gut wall integrity has been identified as a key feature in protecting the body against potentially harmful compounds such as bacteria, toxins and antigens. The gut barrier consists of the mucus barrier, antimicrobial peptides, secretory IgA, the epithelial barrier, and the gut immune system. Gut permeability is reported to increase in sepsis and to play a key role in the development of multi-organ dysfunction. Therefore, gut permeability markers might have the potential to predict the risk of progression from sepsis to severe sepsis. The mechanisms leading to increased gut permeability are not completely clear, yet. Direct and indirect interactions of pathogens, hormonal imbalances, beta-adrenergic activity, hyperglycemia and cytokine activation as well as individual predisposition have been proposed. It seems that increased gut permeability is the common final pathway of a multitude of influencing factors.

Furthermore, the importance of gut microbiota composition has recently been recognized in several diseases; however, not much is known about the role of the microbiome in sepsis to date. Available data suggest, that disturbances in microbiome homeostasis are present in sepsis, but it is yet unknown if these changes are cause or consequence of sepsis. Changes in gut barrier and/or gut microbiota can lead to an increase in microbial products in circulation, contributing to (inadequate) activation and later "paralysis" of immune cells. It is not yet known if the gut microbiome of a patient in early stages of sepsis differs from the healthy microbiome or from the microbiome of a patient in late stages of sepsis. Also, the possibility to modulate the gut microbiome in early sepsis has not been studied yet.

A typical strategy to modulate the gut microbiome is the use of probiotic bacteria. In sepsis, the use of probiotics is well established for specific indications, such as necrotising enterocolitis in neonates, however, studies in adults are scarce. Therefore the aim of this study is to investigate if the ingestion of a multispecies probiotic in early sepsis is able to modulate gut microbiota and/or gut permeability and observe the clinical outcome of treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Age above 18 years
* Sepsis as defined by the presence of a systemic inflammatory response syndrome (2 out of the four: elevated heart rate (tachycardia) >90 beats per minute at rest; body temperature either high (>100.4 F or 38 C) or low (<96.8 F or 36 C); increased respiratory rate of >20 breaths per minute or a reduced partial pressure of carbon dioxide (PaCO2) in arterial blood level; abnormal white blood cell count (>12,000 cells/µL or <4,000 cells/µL or >10% bands [an immature type of white blood cell]) and a known or suspected infection
* Blood cultures ordered by the attending physician

Exclusion Criteria:

* Severe sepsis or septic shock as defined by the Surviving Sepsis Guidelines [1]
* Admission to any intensive care unit or intermediate care unit for any reason
* soluble urokinase plasminogen activator receptor (sUPAR) level at admission >9.15 ng/mL [19]
* Positive beta-D-glycan test
* Patients receiving (par)enteral nutrition
* Presence or suspicion of acute pancreatitis
* Inability to understand and sign an informed consent
* Pregnancy or women of childbearing age without adequate contraception
* Women who are breast-feeding
* Known malignancy or any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | 4 weeks
  next generation sequencing

SECONDARY OUTCOMES:
gut permeability | 4 weeks
  enzyme linked immunosorbent assay
endotoxin | 4 weeks
  limulus amoebocyte assay
soluble sepsis markers | 4 weeks
  enzyme linked immunosorbent assay
neutrophil function | 4 weeks
  flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer-Köllner, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria